CLINICAL TRIAL: NCT06593821
Title: Evaluation of the Effect of Occlusal Splint and Botulinum Toxin Therapies on Masseter Muscle Thickness and Pain Levels on Bruxism Patients
Brief Title: Effect of Different Treatment Techniques on Masseter Muscle Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Şükriye Ece Geduk, Assistant Professor, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/14-4836
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bruxism; Masseter Muscle Hypertrophy
Keywords: Botulinum toxin; Bruxism; Masseter muscle hypertrophy; Occlusal splint; Ultrasound
MeSH Terms: conditions — Bruxism; Masticatory Muscles, Hypertrophy of | interventions — Occlusal Splints; Mouth Protectors; Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control (C) (Experimental): The control group received only preventive recommendations
  Interventions: Behavioral: preventive advice
- Occlusal splint (O) (Experimental): Occlusal splint applied to the upper jaw
  Interventions: Device: Occlusal splint
- Botulinum toxin (B) (Experimental): Botulinum toxin injection applied
  Interventions: Drug: Botulinum toxin
- Occlusal splint and Botulinum toxin (OB) (Experimental): Both occlusal splint and botulinum toxin were applied
  Interventions: Device: Occlusal splint; Drug: Botulinum toxin

INTERVENTIONS:
Device: Occlusal splint — The occlusal splint was fabricated from a 2 mm hard splinting resin material on the plaster model obtained by taking impressions of the patients' upper jaw.
  Other Names: mouthguard
  Arms: Occlusal splint (O); Occlusal splint and Botulinum toxin (OB)
Behavioral: preventive advice — Control group given protective advice such as supporting the jaw when yawning, not chewing gum, not opening the mouth for too long and not opening it too wide, and chewing on both sides when eating.
  Other Names: preventive behaviour
  Arms: Control (C)
Drug: Botulinum toxin — A total of 50 U of botulinum toxin, 25 U in each muscle, was injected
  Other Names: botox
  Arms: Botulinum toxin (B); Occlusal splint and Botulinum toxin (OB)

SUMMARY:
This study aims to evaluate the effects of different treatment techniques on masseter muscle thickness, pain levels and maximum mouth opening in patients with bruxism. The null hypothesis of the study is that there is no difference between the use of an occlusal splint and botulinum toxin on masseter muscle thickness in patients with bruxism.

DETAILED DESCRIPTION:
The study was carried out on 48 patients between 21 and 52 years, who attended the clinic with the complaints of bruxism. The first group was referred to as the Control group (C) and given protective advice such as supporting the jaw when yawning, not chewing gum, not opening the mouth for too long and not opening it too wide, and chewing on both sides when eating. The second group was treated with an occlusal splint (O), the third group with an injection of botulinum toxin (B), and the fourth group with both an occlusal splint and an injection of botulinum toxin (OB). At the beginning of the treatment and after 1, 3 and 6 months, the thickness of the masseter muscles of all patients was measured bilaterally by ultrasound in relaxed and contracted positions. Maximum mouth opening values was recorded by measuring the distance between the incisal edges of the maxillary and mandibular first incisors (teeth 11 and 41) using calipers. Pain levels were assessed using the Visual Analogue Scale (VAS), where patients marked their pain severity on a 10 cm unmarked straight line, with scores ranging from 0 to 10.

Ultrasound measurements Masseter muscle thickness measurements were performed by the same radiologist, using a MyLabTMTwice ultrasound device equipped with a linear probe with a frequency range of 4-13 megahertz. To ensure reproducibility, the probe was positioned perpendicular to the ramus, aligned with the imaginary line between the corner of the lip and the inferior border of the tragus. Measurements were taken at the thickest part of the masseter muscle, with bilateral assessments in both the relaxed and contracted states.

Application of the occlusal splint The occlusal splint was fabricated from a 2 mm hard splinting resin material on the plaster model obtained by taking impressions of the patient's upper jaw. Centric and eccentric occlusal relationships were assessed to ensure equal contact between all teeth. Patients were instructed to wear the splint overnight for at least 8 hours. Patients were also educated on the care and maintenance of the splint and compliance was checked at follow-up visits.

Botulinum toxin injection All injections were administered by the same specialist maxillofacial surgeon. For each dose of 1.0 U/0.1 mL, 100 U of lyophilized botulinum toxin was diluted with 2 cc of saline. The skin area was cleansed with povidone iodine and dried. The anterior, posterior, superior and inferior borders of the masseter muscle were marked to ensure safe injection. Before injection, patients were instructed to clench their teeth to make the injection sites more visible. Intramuscular injections were performed with the needle perpendicular to the skin. A total of 50 U of botulinum toxin was injected , 25 U in each muscle, using 30-gauge injectors.

ELIGIBILITY:
Inclusion Criteria:

* Who volunteered to participate in the study,
* Eighteen years of age or older,
* Has not received any treatment for bruxism before,
* Systemically healthy,
* Visible tooth wear,
* History of clenching or grinding with masticatory pain,
* Morning temporomandibular joint (TMJ) stiffness,
* Masseter hypertrophy

Exclusion Criteria:

* Systemic disease,
* Under the age of eighteen,
* Having received any pharmacological, dental, etc. treatment for bruxism before,
* With any known drug allergy,
* During pregnancy or breastfeeding,
* Bleeding irregularities,
* With mental retardation,
* Active orthodontic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Muscle thickness | 6 months
  Both relaxed and contracted masseter muscle thicknesses were measured by ultrasonography 1, 3 and 6 months after treatment.
Maximum mouth opening | 6 months
  The maximum mouth opening of the patients 1, 3 and 6 months after treatment was recorded by measuring the incisal distance between the upper and lower central incisors.
VAS | 6 months
  Patients were asked to rate their pain levels from 1 to 10 at 1, 3 and 6 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Şükriye E Geduk, Asst. Prof., Study Director — Zonguldak Bulent Ecevit University
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yurttutan ME, Tutunculer Sancak K, Tuzuner AM. Which Treatment Is Effective for Bruxism: Occlusal Splints or Botulinum Toxin? J Oral Maxillofac Surg. 2019 Dec;77(12):2431-2438. doi: 10.1016/j.joms.2019.06.005. Epub 2019 Jun 19. PMID 31302066
- [Background] Lee SJ, McCall WD Jr, Kim YK, Chung SC, Chung JW. Effect of botulinum toxin injection on nocturnal bruxism: a randomized controlled trial. Am J Phys Med Rehabil. 2010 Jan;89(1):16-23. doi: 10.1097/PHM.0b013e3181bc0c78. PMID 19855255
- [Background] Erdil D, Bagis N, Eren H, Camgoz M, Orhan K. The Evaluation of the Relationship between Changes in Masseter Muscle Thickness and Tooth Clenching Habits of Bruxism Patients Treated with Botulinum Toxin A. J Med Ultrasound. 2022 Aug 18;31(1):22-28. doi: 10.4103/jmu.jmu_51_22. eCollection 2023 Jan-Mar. PMID 37180633